CLINICAL TRIAL: NCT01351363
Title: PREDICTION OF POST OPERATIVE PAIN FOLLOWING ARTHROSCOPIC SHOULDER SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Fife (Other Government)
Responsible Party: Doctor Anthony Davis, NHS Fife
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SHLDR1
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Arthroscopic Shoulder Surgery; Pain Threshold
Keywords: Arthroscopic shoulder surgery; Pain threshold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical pain threshold measrement patients (Experimental)
  Interventions: Device: Electrical pain threshold measurement; Device: Measurement of electrical pain threshold

INTERVENTIONS:
Device: Electrical pain threshold measurement — Assessment of preoperative pain threshold using electrical stimulation using a Painmatcher machine.
  Other Names: Pain Matcher ® (Cefar Medical AB, Lund, Sweden)
Device: Measurement of electrical pain threshold — Measurement of preoperative electrical pain threshold and self reporting of postoperative pain scores (for 4 days) on VAS.
  Other Names: Pain Matcher ® (Cefar Medical AB, Lund, Sweden)

SUMMARY:
Following arthroscopic shoulder surgery a small but significant number of people suffer severe postoperative pain.

This study aims to predict which patients are at risk of developing severe post operative pain so that they may be targeted with a more aggressive post operative pain regimen.

DETAILED DESCRIPTION:
Patients presenting for elective (day case) arthroscopic shoulder surgery for either Arthroscopic Subacromial Decompression (ASD Group) or Rotator Cuff Repair (RCR Group) are recruited. Using a Cefar PainMatcher, a pain and sensory threshold assessment tool, consenting patients will have their preoperative pain thresholds recorded. The patients will then have a standard anaesthetic administered with TIVA (propofol/remifentanil) and either a subacromial injection (ASD Group) or interscalene block (RCR Group). Four days following surgery a telephone questionnaire will be completed by the patients recording their worst pain score since surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older able to give informed consent undergoing arthroscopic shoulder surgery at NHS Fife (ASD or rotator cuff repair)

Exclusion Criteria:

* Unable to give informed consent
* Allergy to remifentanil, propofol or levobupivacaine.
* Absence of contralateral arm (thumb/fingers)
* Documented sensory abnormality (e.g. peripheral neuropathy)
* Those not consenting to subacromial injection or interscalene block intraopertively (part of routine management after surgery).
* Psychiatric disease (documented history in Hospital notes or GP referral summary)
* Drug or alcohol misuse (suspicion of or documented)
* No telephone or unable to communicate in English (no interpreter service available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Post operative pain level | 4 days
  Post operative pain level recorded on a VAS (0-10) at rest and movement for the first four days pots shoulder surgery. This information will be correlated with the preoperative pain threshold of patients taken with the Pain matcher machine.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Davis, MBChB, Principal Investigator — NHS Fife
Locations (1):
- Victoria Hospital, Kirkcaldy, Fife, United Kingdom

REFERENCES:
- [Derived] Davis A, Chinn DJ, Sharma S. Prediction of post-operative pain following arthroscopic subacromial decompression surgery: an observational study. F1000Res. 2013 Feb 4;2:31. doi: 10.12688/f1000research.2-31.v1. eCollection 2013. PMID 24358863